CLINICAL TRIAL: NCT00900770
Title: Implications of Amyloid Deposition in Clinically Normal Older Individuals
Brief Title: Implications of Amyloid Pathology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Reisa Sperling, MD, Director of Clinical Research, Memory Disorders Unit, Brigham and Women's Hospital
Other Study IDs: IA0158; 2P50AG005134-268381; 2P50AG005134 (NIH)
Record Dates: First submitted 2009-05-11; First posted 2009-05-13 (Estimated); Last update posted 2009-12-29 (Estimated); Status verified 2009-12

CONDITIONS: Alzheimer's Disease
Keywords: dementia; mild cognitive impairment; beta amyloid
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction; Plaque, Amyloid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- PIB+ NC: PIB positive, cognitively normal individuals with foci of elevated PIB retention in cortical regions typically affected in AD
- PIB- NC: PIB negative, cognitively normal individuals without amyloid deposition

SUMMARY:
The purpose of this study is to determine whether asymptomatic older individuals with high amyloid burden will subsequently manifest cognitive impairment and eventually progress to clinical Alzheimer's Disease (AD).

DETAILED DESCRIPTION:
There is compelling evidence supporting amyloid as one of the key pathologic agents in AD. Autopsy studies suggest the amount and location of fibrillar amyloid deposition does not relate strongly to the degree and type of clinical impairment, compared to tau pathology and neuronal loss. A substantial percentage of individuals known to be cognitively intact prior to death demonstrate significant amyloid pathology at autopsy. PIB-PET studies of older normal individuals have also demonstrated significant amyloid deposition in substantial percentages.

This study will test the hypothesis that amyloid is associated with synaptic dysfunction and neuronal damage. While some individuals are able to compensate for amyloid-related toxicity for an extended time period, sensitive imaging and neuropsychological markers will reveal that normal subjects with evidence of high amyloid burden do demonstrate evidence of abnormality consistent with prodromal AD.

The study will use a combination of functional, structural, and cognitive measures to detect early effects of amyloid deposition, and will utilize PIB retention in order to characterize the relationship of amyloid to neuropsychological and imaging markers of prodromal AD. The relationship of PIB retention to genetic, plasma and cerebrospinal fluid (CSF) biomarkers will be explored. These preliminary data will be used to determine whether asymptomatic older individuals with high amyloid burden will subsequently manifest cognitive impairment and eventually progress to clinical AD. When completed, this project will either provide evidence that the presence of amyloid deposition is a useful biomarker for incipient AD or raise the possibility that amyloid deposition examined in isolation is insufficient to predict early symptoms and progression of AD.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 60 to 90 years
* Clinical Dementia Rating (CDR) Score of 0
* Mini Mental State Exam of 27-30
* A study partner who can answer questions pertaining to daily functioning
* Perform within 1.5 standard deviation of age and education matched norms on screening tests of attention and executive function, language, visuospatial perception and episodic memory
* Stable medications for at least 30 days
* Fluent in English
* Modified Hachinski Score of <4
* Geriatric Depression Scale Score <10

Exclusion Criteria:

* Diagnosis of MCI or dementia
* Individuals with contraindications to MRI (i.e., implanted metal including pacemakers, cerebral spinal fluid shunts, aneurysm clips, artificial heart valves, ear implants or metal/foreign objects in the eyes and those with a history of claustrophobia)
* Unstable medications or on medications with CNS effects including cholinesterase inhibitors, memantine, and antidepressants
* Major psychiatric disorders such as schizophrenia, schizoaffective disorder, major affective disorder, or treatment with ECT (mild depression that is well treated with stable dose of SSRI antidepressants will be allowed)
* Multiple sclerosis or other autoimmune disorders
* Huntington's disease
* Head injury, post-traumatic dementia or seizures
* Metabolic encephalopathy, CNS infection, hydrocephalus
* Cardiovascular disease, stroke, congestive heart failure
* Substance abuse within the past 2 years
* Active cancer
* Active hematological, renal, pulmonary, endocrine or hepatic disorders

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Longitudinal cohort of the Massachusetts Alzheimer's Disease Research Center and community volunteers
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-11; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Compound B (PiB) and F-18 fluorodeoxyglucose (FDG) PET Scan | at 1 month

SECONDARY OUTCOMES:
Cognitive and functional assessments | Baseline and annually for 5 years
Lumbar Puncture (optional) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Reisa Sperling, MD, Principal Investigator — Director of Clinical Research, Memory Disorders Unit, Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Dickerson BC, Bakkour A, Salat DH, Feczko E, Pacheco J, Greve DN, Grodstein F, Wright CI, Blacker D, Rosas HD, Sperling RA, Atri A, Growdon JH, Hyman BT, Morris JC, Fischl B, Buckner RL. The cortical signature of Alzheimer's disease: regionally specific cortical thinning relates to symptom severity in very mild to mild AD dementia and is detectable in asymptomatic amyloid-positive individuals. Cereb Cortex. 2009 Mar;19(3):497-510. doi: 10.1093/cercor/bhn113. Epub 2008 Jul 16. PMID 18632739
- [Background] Aizenstein HJ, Nebes RD, Saxton JA, Price JC, Mathis CA, Tsopelas ND, Ziolko SK, James JA, Snitz BE, Houck PR, Bi W, Cohen AD, Lopresti BJ, DeKosky ST, Halligan EM, Klunk WE. Frequent amyloid deposition without significant cognitive impairment among the elderly. Arch Neurol. 2008 Nov;65(11):1509-17. doi: 10.1001/archneur.65.11.1509. PMID 19001171
- [Background] Jack CR Jr, Lowe VJ, Senjem ML, Weigand SD, Kemp BJ, Shiung MM, Knopman DS, Boeve BF, Klunk WE, Mathis CA, Petersen RC. 11C PiB and structural MRI provide complementary information in imaging of Alzheimer's disease and amnestic mild cognitive impairment. Brain. 2008 Mar;131(Pt 3):665-80. doi: 10.1093/brain/awm336. Epub 2008 Feb 7. PMID 18263627
- [Background] Mintun MA, Larossa GN, Sheline YI, Dence CS, Lee SY, Mach RH, Klunk WE, Mathis CA, DeKosky ST, Morris JC. [11C]PIB in a nondemented population: potential antecedent marker of Alzheimer disease. Neurology. 2006 Aug 8;67(3):446-52. doi: 10.1212/01.wnl.0000228230.26044.a4. PMID 16894106